CLINICAL TRIAL: NCT01533987
Title: Effects of Juice Plus+® Supplementation on Endothelial Function in Overweight Men: A Randomized, Controlled Trial
Brief Title: Effects of Juice Plus+® Supplementation on Endothelial Function in Overweight Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Griffin Hospital (Other)
Collaborators: NSA, LLC (Industry)
Responsible Party: David L. Katz, Yale Griffin Prevention Research Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2009-06
Record Dates: First submitted 2011-08-09; First posted 2012-02-16 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2011-08

CONDITIONS: Overweight and Obesity
Keywords: Male; Overweight; Juice Plus
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Juice Plus (Experimental): Juice Plus is the combination of Juice Plus+® Garden Blend, Juice Plus+® Orchard Blend and Juice Plus+® Vineyard Blend.
  Interventions: Dietary Supplement: Juice Plus
- Placebo (Placebo Comparator): The placebo consists of microcrystalline cellulose,dicalcium phosphate, magnesium stearate, and FD & C yellow #6.
  Interventions: Dietary Supplement: Juice Plus

INTERVENTIONS:
Dietary Supplement: Juice Plus — Juice Plus is the combination of Juice Plus+® Garden Blend, Juice Plus+® Orchard Blend and Juice Plus+® Vineyard Blend.

SUMMARY:
The purpose of the study is to determine the effects of daily ingestion of Juice Plus+® capsules containing Orchard, Garden and Vineyard blends on endothelial function and biomarkers of oxidative stress (oxidized LDL, lipid hydroperoxides and protein carbonyls) in overweight men as compared to the placebo group.

DETAILED DESCRIPTION:
The prevalence of obesity in both adults and children in the United States has increased significantly over the past 50 years. More than 66% of adults in the US are now overweight or obese and at least 17% of children in the population at large are now considered overweight. Obesity may be a factor predisposing patients to a myriad of different comorbidities that increase the associated mortality rate. Several large prospective trials have documented that obesity is an independent risk factor for all-cause mortality from cardiovascular disease (CVD). Considering the major metabolic and biochemical changes that occur in obesity, such as atherogenic dyslipidemia, insulin resistance and hyperinsulinemia, endothelial dysfunction, and chronic inflammatory and prothrombotic states, obesity plays a role in the pathogenesis of systemic atherosclerosis and its clinical complications. Antioxidants are thought to help preserve the endothelium's capacity to generate NO, which acts to promote vasodilation, stabilize platelets, and promote the anti-inflammatory abilities of the endothelium. Juice Plus+® Capsules containing Orchard, Garden and Vineyard blends are rich in the traditional antioxidants β-carotene, Vitamin E and Vitamin C along with other carotenoids and phytonutrients. There is increasing attention to the possibility that micronutrients may exert health effects in concert. Outcomes in studies of isolated micronutrients, such as vitamin E, have often been often disappointing. Plant-derived micronutrients have the potential to contribute to vascular health by offering the endothelium protection from oxidative stress. Evidence of this anticipated effect would have implications for strategies to prevent or retard cardiovascular disease. Endothelial function testing using high-frequency ultrasound imaging of the brachial artery to assess endothelium-dependent flow-mediated dilatation (FMD) offers a non-invasive, uniquely valuable means of assessing aggregated influences on cardiac risk by gauging a physiologic response of the vascular endothelium. Proposed, therefore, is a randomized, double-blinded and placebo-controlled clinical trial of Juice Plus+® on endothelial function in overweight men with central adiposity.

ELIGIBILITY:
Inclusion Criteria:

1. Male age 25-75 years
2. Healthy (no known diabetes mellitus, cardiovascular disease, or eating disorder)
3. Non-smoker
4. Overweight (BMI ≥25) with central adiposity as indicated by waist circumference (≥102 cm).
5. Endothelial dysfunction with high-fat meal

Exclusion Criteria:

1. Use of lipid-lowering or antihypertensive medications, unless stable on medication for at least 3 months and willing to refrain from taking medication for 12 hours prior to EF scanning;
2. Regular use of multivitamins and/or complementary or alternative supplement therapy (including all Juice Plus+® products) and unwillingness to discontinue supplementation for at least 8 weeks prior to study initiation and for study duration
3. Anticipated inability to complete or comply with study protocol;
4. Diagnosed eating disorder
5. Any rheumatologic disease requiring regular use of NSAIDs or alternative medications
6. Regular use of fiber supplements
7. Use of insulin, glucose sensitizing medication, or vasoactive medication
8. Substance abuse (chronic alcoholism, or other chemical dependency
9. Pre-existing cardiovascular disease.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | 8 weeks
  Brachial artery flow mediated dilation (FMD)

SECONDARY OUTCOMES:
Weight | 8 weeks
Waist Circumference | 8 weeks
Blood pressure | 8 weeks
Serum biomarker measures | 8 weeks
  These samples will be used to assess participants' biomarkers of oxidative stress (i.e. oxidized LDL levels, lipid hydroperoxides, and protein carbonyls) and compliance measure (i.e. serum carotenoids)

CONTACTS AND LOCATIONS:
Overall Officials: David L Katz, MD, MPH, Principal Investigator — Yale-Griffin Prevention Research Center
Locations (1):
- Yale-Griffin Prevention Research Center, Derby, Connecticut, United States